CLINICAL TRIAL: NCT06353048
Title: Short Term Radiological and Clinical Outcomes of Fixation of Schatzker II Tibial Plateau Fractures by Screws Only Versus Plate and Screws , Comparative Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Diaaeldin Hamouda, Resident of Orthopaedic department, Sohag University Hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-02-04MS
Record Dates: First submitted 2024-03-17; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Tibial Plateau Fractures Schatzker Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): patients with tibial plateau fractures Schatzker type II fixed by screws only
  Interventions: Procedure: fixation of tibial plateau fractures
- group B (Active Comparator): patients with tibial plateau fractures Schatzker type II fixed by plate and screws
  Interventions: Procedure: fixation of tibial plateau fractures

INTERVENTIONS:
Procedure: fixation of tibial plateau fractures — fixation of tibial plateau fractures by screws only versus plate and screws

SUMMARY:
Tibial plateau fractures are complex injuries produced by high- or low-energy trauma. They principally affect young adults or the 'third age' population ,the tibial plateau is a major weight-bearing surface within the largest and most kinematically complex joint in the human body. Fractures occur as a result of a combination of an axial loading force and a coronal plane (varus/valgus) moment leading to articular shear and depression and mechanical axis malalignment,So Limb alignment and articular surface restoration, allowing early knee motion, are the main goals of surgical treatment.

Soft-tissue damage in fractures around the knee is of critical importance. The oedema and inflammation associated with the trauma can easily lead to local venous compromise, dermal hypoxia, and additional soft-tissue injury. This commonly leads to blistering of the skin and in some cases dermal and even muscle necrosis. Blood-filled blisters should be expected to be associated with a worse outcome than clear fluid-filled ones. Management in the early stages of treatment should focus on preventing further soft-tissue injury while waiting to repair the fracture.

Traditionally, initial radiograph diagnosis should include anteroposterior (AP), lateral and oblique views. But single radiographs do not allow an exact fragment identification and the initial fracture classification can change in 5% to 24% (mean 12%) of cases and treatment can change in up to 26% of cases after CT scan imaging . These findings and the wider availability of CT scanning have made the oblique views less important in the diagnosis. Intra- and peri-articular soft-tissue structures can be affected even in less complex fracture patterns and some X-ray or CT scan data can also suggest the existence of a lateral or medial meniscal tear. Articular depression > 6 mm and/or articular widening > 5 mm are associated with the existence of lateral meniscus, lateral collateral ligament (LCL) or posterior cruciate ligament injuries .

Schatzer classification (published in 1974) will be used to complete understanding of the personality of these fracture which is the key element in decision making process when choosing the best possible treatment .

In general ,tibial plateau fracture are to be operated on , but the decision whether to be operated or not on a specific fracture should be based on the fracture morphology ,soft tissues , the patient general condition and the expected limb axis and articular surface restoration.

Usual indications for surgical treatment are :

1. Intra-articular displacement of ⩾ 2 mm
2. Metaphyseal -diaphyseal translation > 1 cm
3. Angular deformity more than 10 degree in the coronal or sagittal view
4. Open fracture , compartment syndrome and associated ligament injury require repair.
5. Associated fractures of the ipsilateral tibia or fibula

Frequently the depressed articular fragments have to elevated back toward the knee , followed by fixation and sometimes supplemented with bone graft to fill any cancellous bone voids left beneath the joint surface after fracture reduction .

We will evaluate treatment outcomes of closed reduction and percutaneous cannulated screw fixation for tibial plateau fractures versus open reduction and fixation by plate

ELIGIBILITY:
Inclusion Criteria:

* skeletally mature patients aging 18 to 70 years .
* Patient with type II (split depression of lateral tibial plateau )

Exclusion Criteria:

* Severe comminution with >5 mm depression,
* Open fractures,

  * Compartment syndrome, or
* Vascular injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
range of motion of knee joint using Rasmussen score | 1 year
  The primary oucome that we like to measure is range of motion of knee joint on flexion and extension of the joint .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Prat-Fabregat S, Camacho-Carrasco P. Treatment strategy for tibial plateau fractures: an update. EFORT Open Rev. 2017 Mar 13;1(5):225-232. doi: 10.1302/2058-5241.1.000031. eCollection 2016 May. PMID 28461952
- [Background] Salduz A, Birisik F, Polat G, Bekler B, Bozdag E, Kilicoglu O. The effect of screw thread length on initial stability of Schatzker type 1 tibial plateau fracture fixation: a biomechanical study. J Orthop Surg Res. 2016 Nov 22;11(1):146. doi: 10.1186/s13018-016-0484-9. PMID 27876042
- [Background] Giordano CP, Koval KJ, Zuckerman JD, Desai P. Fracture blisters. Clin Orthop Relat Res. 1994 Oct;(307):214-21. PMID 7924035
- [Background] Chan PS, Klimkiewicz JJ, Luchetti WT, Esterhai JL, Kneeland JB, Dalinka MK, Heppenstall RB. Impact of CT scan on treatment plan and fracture classification of tibial plateau fractures. J Orthop Trauma. 1997 Oct;11(7):484-9. doi: 10.1097/00005131-199710000-00005. PMID 9334949